CLINICAL TRIAL: NCT02852161
Title: The Accuracy and Acceptability of Magnet Assisted Capsule Endoscopy in the Diagnosis of Esophageal Pathology: a Pilot Study
Acronym: MACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15109
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Barrett's Oesophagus; Oesophageal Varices
MeSH Terms: conditions — Barrett Esophagus; Esophageal and Gastric Varices | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MACE (Experimental): MACE procedure
  Interventions: Device: Magnet assissted capsule endoscopy
- OGD (Active Comparator): Clinically indicated gastroscopy
  Interventions: Device: Magnet assissted capsule endoscopy

INTERVENTIONS:
Device: Magnet assissted capsule endoscopy — Patients due to have a clinically indicated gastroscopy will be asked to have a MACE procedure on the same day

SUMMARY:
A pilot study to assess the accuracy and acceptability of a magnet assisted capsule endoscopy in detecting esophageal pathology compared to standard endoscopy.

DETAILED DESCRIPTION:
This will be a single centre feasibility study performed at Nottingham University Hospitals NHS Trusts.

We will assess the accuracy of MACE compared to gastroscopy in diagnosing Barretts oesophagus and esophageal varices. Patients will have both tests on the same ay, with the endoscopic findings compared.

ELIGIBILITY:
Inclusion Criteria:

Due to have a clinically indicated gastroscopy Barrett's oesophagus/ oesophageal varices or Controls Able to give informed consent

Exclusion Criteria:

Unable to give consent Pregnant Pacemaker swallowing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuarcy | immediate
  endoscopic

SECONDARY OUTCOMES:
comfort | 2 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Krish Ragunath, Study Chair — Nottingham University
Locations (1):
- Nottingham University Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beg S, Card T, Warburton S, Rahman I, Wilkes E, White J, Ragunath K. Diagnosis of Barrett's esophagus and esophageal varices using a magnetically assisted capsule endoscopy system. Gastrointest Endosc. 2020 Apr;91(4):773-781.e1. doi: 10.1016/j.gie.2019.10.031. Epub 2019 Oct 31. PMID 31678203